

KYOWA Kirin Pharmaceutical Development, Inc 6002-018

### Statistical Analysis Plan

A Phase 3, Long-term, Open-label Study of Istradefylline in Subjects with Moderate to Severe Parkinson's Disease

Protocol Number: 6002-018

US IND Number: 58,356 EudraCT Number: 2015-003887-34

Date: 21 June 2017

#### **Confidentiality Statement**

The information contained in this document is the property of or under the control of Kyowa Kirin Pharmaceutical Development, Inc. and its affiliated companies. This information is provided to you in confidence as an investigator, potential investigator or consultant, for review by you, your staff and applicable Institutional Review Board/Ethics Committee. You shall not disclose this information to others without prior written authorization from Kyowa Kirin Pharmaceutical Development, Inc., except to the extent necessary to obtain informed consent from those persons to whom the drug may be administered, and except as may be required by federal, state, or local laws or regulations.



KYOWA Kirin Pharmaceutical Development, Inc 6002-018

# **Statistical Analysis Plan Signature Page**

| Manager, Biostatistics | Jed Henke | | |
|---|---|---|---|
| Inventiv Health | | Signature | _ |
| | | Date | |
| · · | Junfang) Li PhD | | |
| Kyowa Kırın Pharm<br>212 Carnegie Cente<br>Princeton, NJ 0854<br>Phone: 609-580-571 | 0 | Signature | _ |
| | | Date | |





# Contents

| STAT | FISTICAL ANALYSIS PLAN SIGNATURE PAGE | 2 |
|--------|------------------------------------------------|----|
| LIST | OF ABBREVIATIONS | 5 |
| 1 | INTRODUCTION | 6 |
| 2 | STUDY OBJECTIVES | 7 |
| 2.1 | Primary Objective | 7 |
| 3 | STATISTICAL CONSIDERATIONS OF PROTOCOL | 8 |
| 3.1 | General Statistical Consideration | 8 |
| 3.2 | Overall Study Design and Plan | 8 |
| 3.3 | Treatment Plan | 9 |
| 3.4 | Determination of Sample Size | 10 |
| 3.5 | Disposition of Subjects | 10 |
| 3.6 | Analysis Populations | 10 |
| 3.7 | Demographic and Other Baseline Characteristics | 10 |
| 3.7.1 | Medical History | 11 |
| 3.8 | Prior/Concomitant Medications | 11 |
| 3.9 | Duration of Therapy and Drug Compliance | 11 |
| 3.10 | Efficacy Analysis | 12 |
| 3.11 | Safety Analysis | 12 |
| 3.11.1 | 1 Adverse Events | 13 |
| 3.11.2 | 2 Clinical Laboratory Evaluation | 13 |
| 3.11.3 | Wital Signs, Height and Weight | 14 |
| 3.11.4 | 4 12-Lead Electrocardiogram | 14 |
| 3.11.5 | Physical and Neurological Examinations | 14 |
| 4 | REFERENCES | 15 |
| 5 | PROGRAMMING CONSIDERATIONS | 16 |
| 5.1 | Table, Listing, and Figure Format | 16 |
| 5.1.1 | General | 16 |
| 5.1.2 | Headers | 16 |
| 5.1.3 | Display Titles | 16 |
| 5.1.4 | Column Headers | 17 |



KYOWA Kirin Pharmaceutical Development, Inc 6002-018

| 6 | LIST OF TABLES, LISTINGS, AND FIGURES | 21 |
|-------|-------------------------------------------|----|
| 5.2.5 | Safety | 20 |
| 5.2.4 | Change from Baseline | 20 |
| 5.2.3 | Prior and Concomitant Medications | 20 |
| 5.2.2 | Demographics and Baseline Characteristics | 19 |
| 5.2.1 | Visits | 19 |
| 5.2 | Data-Handling Rules | 19 |
| 5.1.6 | Footnotes | 18 |
| 5.1.5 | Body of the Data Display | 17 |



KYOWA Kirin Pharmaceutical Development, Inc 6002-018

### **List of Abbreviations**

#### **Abbreviations**

AE adverse event

ATC anatomical therapeutic chemical

BP blood pressure
CS clinically significant
ECG electrocardiogram

eCRF electronic case report form

HR heart rate

ICH International Conference on Harmonization
MedDRA Medical Dictionary for Regulatory Activities
PGI-I Patient Global Impression-Improvement

PD Parkinson's Disease
PT preferred term
SAE serious adverse event
SAP Statistical Analysis Plan
SD standard deviation
SOC system organ class

TEAE treatment-emergent adverse event

TLFs tables, data listings, figures

US United States

WHO World Health Organization



KYOWA Kirin Pharmaceutical Development, Inc 6002-018

### 1 INTRODUCTION

This Statistical Analysis Plan (SAP) has been developed after review of Kyowa Kirin Pharmaceutical Development Inc. Protocol 6002-018(final version dated 28 SEP 2015).

This is a Phase 3, 52-week, open-label, flexible-dose, multinational, multicenter study to evaluate the safety and tolerability of istradefylline 20 to 40 mg/d in subjects with moderate to severe Parkinson's Disease (PD) with motor fluctuations and dyskinesia on levodopa combination (levodopa/carbidopa or levodopa/benserazide) therapy plus at least one adjunctive PD medication. For subjects who completed 12 weeks of double-blind treatment and the 30-day follow-up period in Study No. 6002-014, the final study evaluations at Week 12 will serve as the screening evaluations for eligibility for the study. Eligible subjects will initially be treated with istradefylline at a starting dose of 20 mg/d with an option for a dose adjustment to 40 mg/d at Week 12 based on the Investigator's judgment of each subject's response and tolerability. If deemed necessary, one unscheduled dose adjustment visit between Week 2 to Week 12 is allowed in accordance with clinical judgment of the Investigator. Subjects who had a dose adjustment to 40 mg/d can have their dose decreased to 20 mg/d by the Investigator at a second unscheduled dose adjustment visit if there are tolerability issues. The istradefylline dose should remain fixed between Week 26 to Week 52.

This SAP is being written with consideration of the recommendations outlined in the International Conference on Harmonisation (ICH) E9 Guideline entitled "Guidance for Industry: Statistical Principles for Clinical Trials" (ICH Harmonised Tripartite Guideline E9 5FEB1998) and the most recent ICH E3 Guideline entitled, "Guidance for Industry: Structure and Content of Clinical Study Reports" (ICH Harmonised Tripartite Guideline E3 30NOV1995).



KYOWA Kirin Pharmaceutical Development, Inc 6002-018

# **2 STUDY OBJECTIVES**

The objectives of this study are as follows:

# 2.1 Primary Objective

The primary objective of the study is to evaluate the long-term safety and tolerability of oral istradefylline (20 to 40 mg/d) as treatment for subjects with moderate to severe PD.



KYOWA Kirin Pharmaceutical Development, Inc 6002-018

### 3 STATISTICAL CONSIDERATIONS OF PROTOCOL

#### 3.1 General Statistical Consideration

Descriptive statistics (number of subjects, mean, standard deviation [SD], median, minimum, and maximum) for continuous variables and frequency distributions and percentages for discrete (or any categorical) variables will be utilized. The mean and median values will be displayed to one decimal place greater than the original value and the measure of variability (i.e., SD) will be displayed to two decimal places greater than the original value. All summaries and analyses conducted will be by assigned therapy and/or combined total subjects. The last pre-administration observation will be used as the baseline value for calculating post-administration changes from baseline.

All tabulations of summary statistics, graphical presentations, and statistical analyses will be performed using SAS® Version 9.4 or higher.

# 3.2 Overall Study Design and Plan

This is a Phase III, 52-week, open-label, flexible-dose, multinational, multicenter study to evaluate the safety and tolerability of istradefylline 20 or 40 mg/d in subjects with moderate to severe PD with motor fluctuations and dyskinesia. Evaluations will occur on levodopa combination (levodopa/carbidopa or levodopa/benserazide) therapy plus at least one adjunctive PD medication.

Safety outcomes will be assessed by summary of Adverse Events (AEs) and clinical laboratory tests. Vital signs including blood pressure, heart rate, temperature, respiration, weight, and height will be assessed at Screening. Concomitant medications and adverse events, Patient Global Impression-Improvement (PGI-I), will be assessed at every visit throughout the study. Decrease in the dosages of levodopa combinations (levodopa/carbidopa or benserazide/levodopa) due to levodopa-related events will be permitted at the Investigator's discretion and the extent of levodopa/carbidopa or benserazide/levodopa dose reduction will be captured.

The scheduled study visits and procedures are shown in Table 3.2-1



KYOWA Kirin Pharmaceutical Development, Inc 6002-018

Table 3.2-1 Schedule of Visits

| | | | Open-Label Treatment | | Follow-up<br>30 days | |
|---|---|---|---|---|---|---|
| Procedure | Screening <sup>a</sup> Week -1 (Day -1 to 7) | Baseline<br>Day 1 | Week 12<br>(Day 85<br>± 4 days) | Week 26<br>(Day 183<br>± 4 days) | Week 52<br>or ET<br>(Day 365 ±<br>4 days) | following<br>Week<br>52/ET<br>(± 7 days) |
| Written informed consent | X | | | | | |
| Inclusion/Exclusion criteria | X | | | | | |
| Medical history/Demographics | X | | | | | |
| Physical examination | X | | | | | |
| Weight | X | | | | | |
| Height | X | | | | | |
| Vital signs <sup>b</sup> | X | | | | | |
| Clinical laboratory tests | X | | | X | X | |
| Serum pregnancy test <sup>c</sup> | X | X <sup>d</sup> | X <sup>d</sup> | X | X | |
| Serum FSH <sup>e</sup> | X | | | | | |
| 12-lead ECG | X | | | | | |
| Concomitant medications | X | X | X | X | X | $X^f$ |
| Adverse Events <sup>g</sup> | X | X | X | X | X | $X^f$ |
| PGI-I | X | X <sup>h</sup> | X | X | X | |
| Treatment compliance | | | X | X | X | |
| Dispense study drug | | X | X | X | | |

Note: Visits should occur in the ON state. If possible, subjects should have each visit scheduled for approximately the same time of day from Baseline and onwards.

- b: Vital signs to be measured are blood pressure, heart rate, temperature, and respiration rate; all measurements are to be taken in the ON state.
- c: For women of childbearing potential.
- d: A urine dipstick pregnancy test will be conducted at Baseline and Week 12.
- e: For post-menopausal women only.
- f: Subjects will be contacted by telephone for a follow-up visit 30 days (± 7 days) after their last dose of istradefylline.
- g: If there are tolerability issues, subjects can be seen at an unscheduled visit in accordance with clinical judgment of the Investigator. At these visits, assessments will include concomitant medications, adverse events, and treatment compliance. h: Identification only the "key symptom" on the PGI-I for subjects.
- ECG=electrocardiogra m; ET=Early Termination; FSH=follicle stimulating hormone; PGI-I=Patient Global Impression Improvement Scale

#### 3.3 Treatment Plan

All subjects will be treated with istradefylline at a starting dose of 20 mg/d with an option for a dose adjustment to 40 mg/d at Week 12 based on the Investigator's judgment of each subject's response and tolerability. If deemed necessary, one unscheduled dose adjustment visit between Week 2 to Week 12 is allowed in accordance with clinical judgment of the Investigator. Subjects who had a dose adjustment to 40 mg/d can have their dose decreased to

a: For subjects who have completed 12 weeks of double-blind treatment and the 30-day follow-up period in Study No. 6002-014 immediately prior to entering this study, the Screening Visit for those subjects will correspond to the Follow-up visit of Study No. 6002-014.



KYOWA Kirin Pharmaceutical Development, Inc 6002-018

20 mg/d by the Investigator at a second unscheduled dose adjustment visit if there are tolerability issues. The istradefylline dose should remain fixed between Week 26 to Week 52.

In general, summary tables will display one total column. Subjects with dose adjustments will not be displayed separately except where specified.

### 3.4 Determination of Sample Size

Approximately 300 subjects are anticipated to participate in this study. The sample size was estimated based on the number of subjects anticipated to complete 12 weeks of treatment in Study No. 6002-014 and, of these, the estimated proportion meeting the inclusion/exclusion of this study protocol and the estimated number of eligible subjects who agree to participate.

### 3.5 Disposition of Subjects

Subject disposition will be based on all subjects who are eligible for this study. The number entered, completed, and number discontinuing at each visit will be presented. A summary of reasons for early discontinuation will be provided. Reasons for early discontinuation include AEs, lack of efficacy, protocol violation, or non-compliance with study drug, subject's withdrawal of consent, or other (to be specified by the Investigator).

# 3.6 Analysis Populations

The following analysis populations will be used in the study:

- Intent-to-Treat Set (ITT): Includes all subjects with both a valid screening and at least one valid post-screening efficacy assessment.
- Safety Analysis Set: Includes all subjects who received at least one dose of assigned study drug (even a partial dose).

The number of subjects in each of the ITT and Safety Analysis sets will be presented.

### 3.7 Demographic and Other Baseline Characteristics

Demographic and Baseline characteristics will be summarized descriptively for the ITT and Safety Analysis Sets for each treatment arm and in total. These summaries will include demographics (including age, race, sex, height, weight, daily caffeine intake, smoking status, and body mass index (BMI), medical history, and physical examination results of note. Baseline will be defined as the last observation obtained prior to the first dose of study drug in this study.

All demographic data and Baseline disease characteristics data will be listed by subject.



KYOWA Kirin Pharmaceutical Development, Inc 6002-018

# 3.7.1 Medical History

Medical history for those subjects reporting any past or present conditions at screening will be summarized by body system for the Safety Analysis Set for each treatment arm and in total. Medical history data will be listed by subject.

#### 3.8 Prior/Concomitant Medications

All prior and concomitant medications will be coded to preferred drug names and therapeutic drug class using the World Health Organization (WHO) Drug Dictionary. Prior medications refer to medications taken within 30 days prior to the first dose of study medication (i.e. the duration when taken overlaps the time interval between first dose date minus 30 to first dose date minus 1 at any single time). Concomitant medications are those with start date on or after the date of the first dose or that started prior to the date of the first dose but are indicated as continuing into the treatment period. Any medications with partial start and/or stop dates will be considered concomitant if the assignment is uncertain.

The number and percentage of subjects taking concomitant medications during the treatment period will be summarized by anatomical therapeutic chemical (ATC) and preferred term (PT) for the Safety Analysis Set. If a subject took a coded medication more than once, the subject will be counted once for that coded medication total. If a subject had more than one coded medication in a therapeutic class, the subject will be counted only once in that therapeutic class total.

All prior and concomitant medications will be listed by subject.

### 3.9 Duration of Therapy and Drug Compliance

Duration of therapy will be summarized as the number of weeks [defined as (days from first dosing to last dosing)/7, with precision to one decimal place] receiving treatment from the first day of dosing until the last day of dosing.

The percent compliance for taking study drug as prescribed will be calculated at Weeks 12, 26, and 52 using the formula (with precision to one decimal place):

Compliance over the entire open-label treatment period will be similarly computed using the total number of tablets dispensed from Screening to Week 52 and the total number of tablets returned and the total number of tablets expected to be taken for this period. The number of tablets expected to be taken will be derived as follows: end of study/treatment date minus



KYOWA Kirin Pharmaceutical Development, Inc 6002-018

first treatment date, plus one. If subjects are escalated to 40 mg per day, and are dispensed 20 mg tablets, two tablets per day will be expected and the number of expected tablets for this time period will be derived as follows: end of treatment period date minus first treatment period date, plus one, multiplied by two. Summary statistics for compliance will be presented for the Safety Analysis Set.

Treatment adjustments will be summarized by time period, Baseline to Week 12, >Week 12 to Week 26, and >Week 26 to Week 52. The number of subjects who remained on Istradefylline 20 mg, the number for whom dose was escalated to Istradefylline 40 mg and remained at 40 mg, and the number for whom dose was escalated to Istradefylline 40 mg and later de-escalated to Istradefylline 20 mg will be displayed for each time period.

## 3.10 Efficacy Analysis

All efficacy data collected from the PGI-I scale used in this study will be summarized using descriptive statistics for the ITT population. Summaries will be performed overall and by treatment in 6002-014, Istradefylline versus placebo. The PGI-I scale will be summarized categorically, displaying the number and percentage of subjects in each category outlined below at weeks 12, 26, and 52. PGI-I overall condition score and subscores will be reported (fatigue, sleep, motivated to get tasks done, key symptom).

- 1=Moderate improvement (or greater)
- 2=Mild improvement
- 3=No change from Baseline
- 4=Mild deterioration
- 5=Moderate deterioration (or greater)

No statistical tests (i.e. p-values) will be performed.

### 3.11 Safety Analysis

All safety analyses will be based on the Safety Analysis Set. All continuous safety data collected in this study will be summarized using descriptive statistics at each assessment time based on actual values and change from Baseline values. Baseline is defined as the last non-missing value obtained prior to first treatment. Continuous variables will be summarized using n, mean, SD, median, minimum, and maximum values. Categorical variables will be summarized using the number and percentage of subjects in each category. All out-of-normal-range results and clinically significant changes in any safety variable will be flagged in the subject data listings.



KYOWA Kirin Pharmaceutical Development, Inc 6002-018

#### 3.11.1 Adverse Events

The Medical Dictionary for Regulatory Activities (MedDRA) will be used to classify all AEs reported during the study by system organ class (SOC) and PT. All summary tables will include counts of subjects with treatment-emergent adverse events (TEAEs), defined as those AEs that have a start date after the start of study drug. AEs with missing start dates, but with stop dates either overlapping into the treatment period or missing, will be considered TEAEs, taking the worst-case approach. All other AEs will be classified as non-TEAEs and identified in listings only. An overall summary table of TEAEs will be presented with the number and percentage of subjects having a TEAE, a serious TEAE, a TEAE leading to study discontinuation, a TEAE with an outcome of death, a TEAE related to study drug ('possibly', 'probably', or 'definitely' related), or a severe TEAE. The overall incidence of TEAEs will be summarized by SOC and by SOC and PT using the number and percentage of subjects reporting an event and by the number of events reported. The incidence of TEAEs resulting in death, serious TEAEs, and TEAEs leading to study discontinuation will be summarized in a similar manner. TEAEs will also be summarized by maximum severity (mild, moderate, or severe), and closest relationship to study drug (related or not related) with the percentage of subjects in each category. A TEAE with missing severity or relationship will be considered severe or related, respectively. If more than one TEAE is recorded for a subject within any SOC or PT, the subject will only be counted once within that SOC or PT total. Serious TEAEs, TEAEs leading to study discontinuation, and TEAEs with an outcome of death will also be presented in separate listings.

A summary of TEAEs and drug related TEAEs will be provided by dose at the first occurrence (Istradefyline 20 mg or 40 mg) and by SOC and PT. For subjects uptitrating from 20 mg to 40 mg or down-titrating from 40 mg to 20 mg, treatment start and stop dates will be used to identify the dose level at the time of the event. Subjects receiving both dose levels will be included in the denominator of both dose levels.

### 3.11.2 Clinical Laboratory Evaluation

Actual values and change from Baseline values for continuous data from clinical laboratory tests will be summarized descriptively at all scheduled study. Categorical data from clinical laboratory tests will be similarly summarized for the actual values. Clinical laboratory tests categorized as in or out of normal range will be summarized using shift tables by visit. Shift tables will be the cross tabulation of the Baseline result category (high, normal, low) with post-Baseline result category (high, normal, low) for each visit during the treatment period. All out-of-normal range results will be flagged in the subject data listings.



KYOWA Kirin Pharmaceutical Development, Inc 6002-018

# 3.11.3 Vital Signs, Height and Weight

Vital signs measurements, including heart rate (HR), systolic and diastolic blood pressure (BP), respiratory rate, temperature, height and body weight are collected at screening and will be listed by subject.

### 3.11.4 12-Lead Electrocardiogram

Electrocardiogram (ECG) interpretations by the Investigator are collected at screening and at unscheduled visits based on clinical indication. All ECG overall interpretations will be listed by subject.

### 3.11.5 Physical and Neurological Examinations

Physical and neurological examinations are performed at screening and at unscheduled visits as clinically indicated. All examination findings, including general appearance, head (eyes, ears, nose, and throat), cardiovascular, respiratory, abdominal, musculoskeletal, extremities, lymph nodes, skin, and neurological examination results (cranial nerves, sensory, motor, stance/gait, reflexes, mental status), will be listed by subject.



KYOWA Kirin Pharmaceutical Development, Inc 6002-018

### 4 REFERENCES

- 1. International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use, ICH Harmonised Tripartite Guideline, Statistical Principles for Clinical Trials (E9), 5 February 1998.
- 2. International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use, ICH Harmonised Tripartite Guideline, Structure and Content of Clinical Study Reports (E3), 30 November 1995.



KYOWA Kirin Pharmaceutical Development, Inc 6002-018

### 5 PROGRAMMING CONSIDERATIONS

All tables, data listings, figures (TLFs), and statistical analyses will be generated using SAS® Version 9.4. Generated outputs will adhere to the following specifications.

### 5.1 Table, Listing, and Figure Format

#### 5.1.1 General

- 1) All TLFs will be produced in landscape format.
- 2) All TLFs will be produced using the Courier New font, size 10.
- 3) The data displays for all TLFs will have a 1.5-inch binding margin on top of a landscape oriented page and a minimum 1-inch margin on the other 3 sides.
- 4) Headers and footers for figures will be in Courier New font, size 8.
- 5) Legends will be used for all figures with more than 1 variable, group, or item displayed.
- 6) TLFs will be in black and white (no color).
- 7) Specialized text styles, such as bolding, italics, borders, shading, and superscripted and subscripted text, will not be used in the TLFs. On some occasions, superscripts 1, 2, or 3 may be used (see below).
- 8) Only standard keyboard characters will be used in the TLFs. Special characters, such as non-printable control characters, printer-specific, or font-specific characters, will not be used. Hexadecimal-derived characters will be used, where possible, if they are appropriate to help display math symbols (e.g., µ). Certain superscripts (e.g., cm²) will be employed on a case-by-case basis.
- 9) Mixed case will be used for all titles, footnotes, column headers, and programmer-supplied formats.

#### 5.1.2 Headers

1) All output should have the following header at the top of the page:

Kyowa Kirin Pharmaceutical Development, Inc. Istradefylline: Protocol 6002-018

DDMMMYYYY Page n of N

All output should have page numbers. TLFs should be internally paginated in relation to the total length (i.e., the page number should appear sequentially as page n of N, where N is the total number of pages in the table).

### 5.1.3 Display Titles

1) Each TLF should be identified by a numeral, and the designation (i.e., Table 1) should be centered above the title. A decimal system (14.x.y.z and 16.2.x.y) should be



KYOWA Kirin Pharmaceutical Development, Inc 6002-018

used to identify TLFs with related contents. The title is centered in initial capital characters. The analysis set should be identified on the line immediately following the title. The title and table designation are single spaced. A solid line spanning the margins will separate the display titles from the column headers. There will be 1 blank line between the last title and the solid line.

Table 14.x.y.z
First Line of Title
Second Line of Title if Needed
Analysis Set

#### 5.1.4 Column Headers

- 1) Column headings should be displayed immediately below the solid line described above in initial upper-case characters.
- 2) For numeric variables, include "unit" in column or row heading when appropriate.
- 3) Analysis set sizes will be presented for each treatment group in the column heading as (N=xx) (or in the row headings if applicable). This is distinct from the 'n' used for the descriptive statistics representing the number of subjects in the analysis set.
- 4) The majority of the tables will be summarized using a "Total" column. For those tables displaying "by treatment", the order of treatments will be: Istradefylline 20 mg/day, Istradefylline 40 mg/day, and Total.

# 5.1.5 Body of the Data Display

- 1) Listings will be sorted for presentation in order of treatment groups as above, subject identification, collection day, and collection time (as applicable).
- 2) If the categories of a parameter are ordered, then all categories between the maximum and minimum category should be presented in the table, even if n=0 for all treatment groups in a given category that is between the minimum and maximum level for that parameter. For example, the frequency distribution for symptom severity would appear as:

| Severity Rating | n |
|-----------------|---|
| severe | 0 |
| moderate | 8 |
| mild | 3 |

Where percentages are presented in these tables, any counts of 0 will be presented as 0 and not as 0 (0%).

- 3) If the categories are not ordered (e.g., Medical History, Reasons for Discontinuation from the Study, etc.), then only those categories for which there is at least 1 subject represented in 1 or more groups should be included. Exception, if 'other' category is present with at least 1 subject, all pre-specified categories will be included.
- 4) An Unknown or Missing category for categorical summarization should be added to any parameter for which information is not available for 1 or more subjects.



KYOWA Kirin Pharmaceutical Development, Inc 6002-018

5) Unless otherwise specified, the estimated mean and median for a set of values should be printed out to 1 more significant digit than the original values, and standard deviations should be printed out to 2 more significant digits than the original values. The minimum and maximum should report the same significant digits as the original values. For example, for systolic BP:

| N | XX |
|--------|------------|
| Mean | XXX.X |
| SD | X.XX |
| Median | XXX.X |
| Range | (XXX, XXX) |

- 6) Data in columns of a table should be formatted as follows:
  - alpha-numeric values are left-justified;
  - whole numbers (e.g., counts) are right-justified; and
  - numbers containing fractional portions are decimal aligned.
- 8) Percentage values should be printed with 1 digit to the right of the decimal point in parentheses 1 space after the count (e.g., 7 (12.8%), 13 (5.4%)). Less-than-signs "<0.1%" should be printed when values are >0.0% and <0.1% (not 0.0%). Unless otherwise noted, for all percentages, the number of subjects in the analysis set for the treatment group who have an observation will be the denominator.
- 9) Tabular display of data for prior / concomitant medications, and all tabular displays of adverse event data should be presented by the body system, drug class, or SOC with the highest occurrence in the active treatment group in decreasing order. Within the body system, drug class and SOC, medical history (by PT), drugs (by ATC1 code), and adverse events (by PT) should be displayed in decreasing order. If incidence for more than 1 term is identical, they should then be sorted alphabetically.
- 10) Missing data should be represented on subject listings as either a hyphen ("-") with a corresponding footnote (" = unknown or not evaluated"), or as "N/A", with the footnote "N/A = not applicable", whichever is appropriate. Missing descriptive statistics or p-values due to non-estimability should be reported as "-".
- 11) Dates should be printed in SAS® DATE9.format ("DDMMMYYYY": 01JUL2000). Missing portions of dates should be represented on subject listings as dashes (--JUL2000). Dates that are missing because they are not applicable for the subject are output as "N/A", unless otherwise specified.
- 12) All observed time values must be presented using a 24-hour clock HH:MM:SS format (e.g., 01:35:45, or 11:26). Time will only be reported if it was measured as part of the study.

#### 5.1.6 Footnotes

1) A solid line spanning the margins will separate the body of the data display from the footnotes.



KYOWA Kirin Pharmaceutical Development, Inc 6002-018

- 2) All footnotes will be left justified with single-line spacing immediately below the solid line underneath the data display.
- 3) Footnotes should always begin with "Note:" if an informational footnote, or asterisks and other non-numeric symbols if an annotated footnote. Each new footnote starts on a new line.
- 4) Footnotes will be present on the page where they are first referenced and thereafter on each page of the table, unless the footnote is specific only to certain pages. Subject specific footnotes should be avoided.
- 5) Footnotes will be used sparingly and must add value to the table, figure, or data listing. If more than 4 footnotes are planned, then a cover page may be used to display footnotes, and only those essential to comprehension of the data will be repeated on each page. Footnotes should not repeat definitions already provided in the SAP.
- 6) The last line of the footnote section will be a standard source line that indicates the data source called in by the program, the name of the program used to produce the data display, and the listing source (i.e., 'Data source: xyzabc.sas7bdat Program source: myprogram.sas Listing source: 16.x.y.z').

# 5.2 Data-Handling Rules

This section describes naming conventions and rules for calculations that would be common to all applicable tables. Some rules specific to a table can be found in the relevant mock-ups.

### **5.2.1** Visits

- 1) Relative Study Day: The first day of treatment is Day 1. A minus (-) sign indicates days prior to the start of treatment (e.g., Day -5 represents 5 days before start of therapy. There is no Day 0.). The relative study day for a specific visit is calculated as (Visit Date Date of First Dose +1).
- 2) Baseline: Evaluation taken on Day 1 or the last available evaluation prior to the first dose of study drug if the former is missing.

# 5.2.2 Demographics and Baseline Characteristics

- Age (if derived) = (Date of informed consent Date of birth + 1) / 365.25 and truncated to complete years.
- Conversion factors and calculations for height, weight, and BMI (with precision to one decimal place):
  - Height (in cm) = height (in inches) \* 2.54
  - Weight (in kg) = weight (in lbs) \* 0.4536
  - BMI  $(kg/m^2)$  = Weight $(kg)/[Height(m)^2]$



KYOWA Kirin Pharmaceutical Development, Inc 6002-018

### 5.2.3 Prior and Concomitant Medications

- 1) Prior and concomitant medications will be coded and classified using the WHODRUG dictionary. The specific dictionary version will be provided in the actual tables/listings. Prior medications refer to medications taken within 30 days prior to the first dose of study medication (i.e. the duration when taken overlaps the time interval between first dose date minus 30 to first dose date minus 1 at any single time). Concomitant medications are those with start date/time on or after the date/time of dosing or that started prior to the date/time of dosing but are indicated as continuing into the treatment period. Any medications with partial start and/or stop dates will be considered concomitant if the assignment is uncertain.
- 2) Medications missing both start and stop dates, or having a start date prior to the last dose of study drug and missing the stop date, or having a stop date after the start of study drug and missing the start date, will be counted as concomitant. When partial dates are present in the data, both a partial start date and/or a partial stop date will be evaluated to determine whether it can be conclusively established that the medication either ended prior to the start of study drug or started after the end of study drug. If the above cannot be conclusively established based on the partial and/or present dates, then the medication will be counted as concomitant.

### 5.2.4 Change from Baseline

Change from Baseline is defined as X-baseline for each X value at Weeks 12, 26, and 52.

## 5.2.5 Safety

- 1) If multiple results (e.g., laboratory test results) are reported at a study visit, then the first available result reported for that visit will be used in that visit summary.
- 2) Adverse events will be coded and classified using MedDRA dictionary. The specific dictionary version will be provided in the actual tables/listings.
- 3) Counting rules for TEAEs: Adverse event tables will include all recorded adverse signs and symptoms, except those with onset or stop dates prior to the first day of study drug. Adverse events with missing start dates, but with stop dates either overlapping into the treatment period or missing, will be counted as treatment-emergent, taking the worst-case approach. Special care will be taken regarding partial dates with similar logic to that of the prior/concomitant medications applied.
- 4) For purposes of flagging individual subject data, laboratory abnormalities are defined as values above or below the normal range.
- 5) Conversion factor for body temperature:

Temperature (in  $^{\circ}$ C) = 5/9 \* (Temperature [in  $^{\circ}$ F]-32), with precision to one decimal place.



# 6 LIST OF TABLES, LISTINGS, AND FIGURES

# **Disposition and Demography Tables**

| Table 14.1.1 | Subject Enrollment by Center |
|---|---|
| Table 14.1.2 | Subject Disposition |
| Table 14.1.3 | Demographic and Baseline Characteristics – Safety Analysis Set |
| Table 14.1.4 | Parkinson's Disease History – Safety Analysis Set |
| Table 14.1.5.1 | Prior Medications (Excluding Antiparkinsonian Medications) – Safety Analysis Set |
| Table 14.1.5.2 | Concomitant Medications (Excluding Antiparkinsonian Medications) – Safety Analysis |
| | Set |
| Table 14.1.6.1 | Prior Antiparkinsonian Medications – Safety Analysis Set |
| Table 14.1.6.2 | Concomitant Antiparkinsonian Medications – Safety Analysis Set |
| Table 14.1.7.1 | Duration of Therapy (weeks) – Safety Analysis Set |
| Table 14.1.7.2 | Compliance Rate – Safety Analysis Set |
| Table 14.1.7.3 | Treatment Adjustments – Safety Analysis Set |

# **Efficacy Tables**

| Table 14.2.1.1 | Patient Global Impression - Improvement by Study Visit - Overall Condition - ITT |
|---|---|
| | Analysis Set |
| Table 14.2.1.2 | Patient Global Impression - Improvement by Study Visit - Fatigue - ITT Analysis Set |
| Table 14.2.1.3 | Patient Global Impression - Improvement by Study Visit - Sleep - ITT Analysis Set |
| Table 14.2.1.4 | Patient Global Impression - Improvement by Study Visit - Motivated to Get Things |
| | Done – ITT Analysis Set |
| Table 14.2.1.5 | Patient Global Impression - Improvement by Study Visit - Key Symptom - ITT |
| | Analysis Set |



KYOWA Kirin Pharmaceutical Development, Inc 6002-018

# **Safety Tables**

| Overall Summary of Treatment-Emergent Adverse Events – Safety Analysis Set |
|---|
| Subjects with Treatment-Emergent Adverse Events by System Organ Class and Preferred |
| Term – Safety Analysis Set |
| Subjects with Treatment-Emergent Adverse Events by System Organ Class, Preferred |
| Term, and Maximum Severity – Safety Analysis Set |
| Subjects with Treatment-Emergent Adverse Events by System Organ Class, Preferred |
| Term, and Relationship to Study Drug – Safety Analysis Set |
| Subjects with Treatment-Emergent Adverse Events Leading to Deathby System Organ |
| Class and Preferred Term – Safety Analysis Set |
| Subjects with Serious Treatment-Emergent Adverse Events by System Organ Class and |
| Preferred Term – Safety Analysis Set |
| Subjects with Treatment-Emergent Adverse Events Leading to Discontinuation from the |
| Study by System Organ Class and Preferred Term – Safety Analysis Set |
| Summary Statistics by Laboratory Test: Hematology – Parameter (unit) — Safety |
| Analysis Set |
| Summary Statistics by Laboratory Test: Blood Chemistry – Parameter (unit) –Safety |
| Analysis Set |
| Summary Statistics by Laboratory Test: Urinalysis – Parameter (unit) –Safety Analysis |
| Set |
| Shift Tables by Laboratory Test: Hematology –Safety Analysis Set |
| Shift Tables by Laboratory Test: Blood Chemistry –Safety Analysis Set |
| Shift Tables by Laboratory Test: Urinalysis – Continuous Parameters Safety Analysis Set |
| Shift Tables by Laboratory Test: Urinalysis – Categorical Parameters Safety Analysis Set |



KYOWA Kirin Pharmaceutical Development, Inc 6002-018

# **Listings**

| Listing 16.2.1.1 | Subject Completion/Discontinuation |
|---|---|
| Listing 16.2.1.2 | Screen Failures |
| Listing 16.2.2.1 | Protocol Deviations |
| Listing 16.2.2.2 | Inclusion/Exclusion Criteria |
| Listing 16.2.3 | Subjects Excluded from Analysis Sets |
| Listing 16.2.4.1 | Demography |
| Listing 16.2.4.2 | Parkinson's Disease History |
| Listing 16.2.4.3 | Medical History |
| Listing 16.2.4.4.1 | Prior Medications (Excluding Antiparkinsonian Medications) |
| Listing 16.2.4.4.2 | Concomitant Medications (Excluding Antiparkinsonian Medications) |
| Listing 16.2.4.5.1 | Prior Antiparkinsonian Medications |
| Listing 16.2.4.5.2 | Concomitant Antiparkinsonian Medications |
| Listing 16.2.5.1 | Study Drug Dosing Record and Compliance |
| Listing 16.2.5.2 | Study Drug Dose Adjustment |
| Listing 16.2.6 | Patient Global Impression - Improvement |
| Listing 16.2.7.1 | Adverse Events |
| Listing 16.2.7.2 | Serious Adverse Events and Deaths |
| Listing 16.2.7.3 | Adverse Events Leading to Discontinuation from the Study |
| Listing 16.2.8.1 | Laboratory Assessments - Hematology |
| Listing 16.2.8.2 | Laboratory Assessments – Blood Chemistry |
| Listing 16.2.8.3 | Laboratory Assessments – Urinalysis |
| Listing 16.2.8.4 | Pregnancy Test |
| Listing 16.2.8.5 | Follicle Stimulating Hormone |
| Listing 16.2.8.6 | Laboratory Assessments - Comments |
| Listing 16.2.9.1 | Vital Signs and Body Weight |
| Listing 16.2.9.2 | 12-Lead Electrocardiogram Report – Qualitative Data by Subject |
| Listing 16.2.9.3 | Physical Examination |
| Listing 16.2.9.4 | Neurological Examination |

Table 14.1.1
Subject Enrollment by Center
Enrolled Subjects

| Center | Investigator | Total |
|--------|--------------|----------------------|
| Number | Name | All Safety[1] ITT[2] |
| 1 | Xxxxxx | xx xx xx |
| | Үуууууу | xx xx xx |

| Total | XX | XX |
|-------|----|----|

<sup>[1]</sup> Safety Analysis Set: Includes all subjects who received at least one dose of assigned study drug (even a partial dose).

Data source: xyzabc.sas7bdat Program source: myprogram.sas Listing source: 16.x.y.z

**NOTE TO PROGRAMMER:** Add source to all tables following the same format.

<sup>[2]</sup> Intent-to-Treat (ITT) set includes all subjects with both a valid baseline and at least one valid post-baseline assessment.

Table 14.1.2 Subject Disposition Enrolled Subjects

| Status | Total |
|-------------------------------------|-----------|
| Randomized | xx (100%) |
| ITT Analysis Set [1] | xx (xx.x) |
| Safety Analysis Set [2] | xx (xx.x) |
| Completed | |
| Week 12 | xx (xx.x) |
| Week 26 | xx (xx.x) |
| Week 52 | xx (xx.x) |
| Completed Treatment Period | xx (xx.x) |
| Discontinued Prematurely | xx (xx.x) |
| Adverse Event | xx (xx.x) |
| Prohibited Concomintant Medication | xx (xx.x) |
| Subject withdrew consent | xx (xx.x) |
| Investigator decision | xx (xx.x) |
| Noncompliance | xx (xx.x) |
| Administrative reasons | xx (xx.x) |
| Pregnancy | xx (xx.x) |
| Subject did not meet entry criteria | xx (xx.x) |
| Other | xx (xx.x) |

<sup>[1]</sup> Intent-to-Treat (ITT) set includes all subjects with both a valid baseline and at least one valid post-baseline assessment.

<sup>[2]</sup> All subjects who received at least one dose of assigned study drug (even a partial dose).

Table 14.1.3

Demographic and Baseline Characteristics
Safety Analysis Set

| | Total |
|-------------------------------------------|-----------|
| Variable | (N=) |
| Age (years) | |
| n | xx |
| Mean | XX.X |
| SD | x.xx |
| Median | XX.X |
| Range | (xx, xx) |
| Gender n (%) | |
| Male | xx (xx.x) |
| Female | xx (xx.x) |
| Race n (%) | |
| White | xx (xx.x) |
| Asian | xx (xx.x) |
| Black | xx (xx.x) |
| American Indian or Alaska Native | xx (xx.x) |
| Native Hawaiian or Other Pacific Islander | xx (xx.x) |
| Other | xx (xx.x) |
| Not Applicable | xx (xx.x) |
| Ethnicity n (%) | |
| Hispanic or Latino | xx (xx.x) |
| Not Hispanic or Latino | xx (xx.x) |

Table 14.1.3

Demographic and Baseline Characteristics
Safety Analysis Set

| | Total |
|-------------|----------|
| Variable | (N=) |
| Height (cm) | |
| n | XX |
| Mean | XX.X |
| SD | X.XX |
| Median | XX.X |
| Range | (xx, xx) |
| Weight (kg) | |
| n | XX |
| Mean | XX.X |
| SD | X.XX |
| Median | XX.X |
| Range | (xx, xx) |
| BMI (kg/m2) | |
| n | xx |
| Mean | xx.x |
| SD | x.xx |
| Median | xx.x |
| Range | (xx, xx) |

Table 14.1.3

Demographic and Baseline Characteristics
Safety Analysis Set

| | Total |
|-------------------------------------------|-----------|
| Variable | (N=) |
| Current Smoker n (%) | |
| Yes | xx (xx.x) |
| No | xx (xx.x) |
| Number of Cigarettes Smoked per Day n (%) | |
| <= 5 cigarettes per day | xx (xx.x) |
| > 5 cigarettes per day | xx (xx.x) |
| Number of Cups (8 Ounces) per Day of | |
| Any Caffeinated Beverage | |
| n | xx |
| Mean | XX.X |
| SD | x.xx |
| Median | XX.X |
| Range | (xx, xx) |

NOTE TO PROGRAMMER: Additional baseline characteristics may be added as needed.

Table 14.1.4
Parkinson's Disease History
Safety Analysis Set

| Variable | Total |
|-------------------------------------------------|-----------|
| Statistics | (N=) |
| Time Since Diagnosis (years) n (%) | |
| < 1 year | xx (xx.x) |
| 1-3 years | xx (xx.x) |
| 4-7 years | xx (xx.x) |
| >= 8 years | xx (xx.x) |
| Time Since Initiation of Levodopa (years) | |
| n | xx |
| Mean | xx.x |
| SD | X.XX |
| Median | XX.X |
| Range | (xx, xx) |
| Time Since Onset of Motor Complications (years) | |
| n | xx |
| Mean | xx.x |
| SD | x.xx |
| Median | XX.X |
| Range | (xx, xx) |

Programming note: The data in this table will be brought forward from the Kyowa 6002-14 Study

Table 14.1.5.1
Prior Medications (Excluding Antiparkinsonian Medications)
Safety Analysis Set

| Therapeutic Class/ | Total |
|-------------------------------------|-----------|
| Preferred Term [1] | (N=) |
| Subjects who took prior medications | xx (xx.x) |
| Therapeutic Class 1 | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) |
| Etc. | xx (xx.x) |

Note: This table includes medications that were taken within 30 days prior to the first dose of Iistradefyline. [1] WHODRUG Dictionary Version 2013 SEP was used for coding.

#### **NOTE TO PROGRAMMER:**

Please present medications in descending order of total frequency by therapeutic class and then by descending order of total frequency of preferred term within the therapeutic class.

Kyowa Kirin Pharmaceutical Development, Inc. Istradefylline: Protocol 6002-018

DDMMMYYYY Page n of N

Statistical Analysis Plan Istradefylline 6002-018

Table 14.1.5.2

Concomitant Medications (Excluding Antiparkinsonian Medications)

Safety Analysis Set

#### **NOTE TO PROGRAMMER:**

Follow the same format as Table 14.1.5.1: Change "Subjects who took prior medications" to: "Subjects who took concomitant medications." Change note to "This table includes medications having a start date on or after the date of the first dose of Istradefyline or with a start date prior to the first dose of Istradefyline and continuing beyond the first dose of Istradefyline.".

Table 14.1.6.1
Prior Antiparkinsonian Medications
Safety Analysis Set

#### **NOTE TO PROGRAMMER:**

Follow the same format as Table 14.1.5.1: Change "Subjects who took prior medications" to: "Subjects who took prior antiparkinsonian medications"

Table 14.1.6.2
Concomitant Antiparkinsonian Medications
Safety Analysis Set

#### **NOTE TO PROGRAMMER:**

Follow the same format as Table 14.1.5.2: Change "Subjects who took concomitant medications" to: "Subjects who took concomitant antiparkinsonian medications."

Table 14.1.7.1
Duration of Therapy (Weeks)
Safety Analysis Set

| | Total |
|---------------------------------------|-----------|
| Statistics | (N=) |
| Duration of Therapy (weeks) [1] n (%) | |
| <=12 | xx (xx.x) |
| >12 to <=26 | xx (xx.x) |
| >26 to <=52 | xx (xx.x) |
| >52 | xx (xx.x) |
| | XX |
| n | XX.X |
| Mean | X.XX |
| SD | XX.X |
| Median | (xx, xx) |
| Range | xx |
| Total Duration (subject weeks) | XX |

<sup>[1]</sup> Duration of therapy = ([Last dose date - First dose date] + 1)/7

Table 14.1.7.2 Compliance Rate Safety Analysis Set

| | Total |
|--------------------------|------------|
| Statistics | (N=) |
| Compliance Rate Category | |
| Treatment Period n (%) | |
| <60% | xx (xx.x%) |
| 60 to 69% | xx (xx.x%) |
| 70 to 79% | xx (xx.x%) |
| 80 to 89% | xx (xx.x%) |
| 90 to 99% | xx (xx.x%) |
| 100 to 109% | xx (xx.x%) |
| >110% | xx (xx.x%) |
| n | xx |
| Mean Rate | XX.X |
| Median Rate | xx.x |
| Week 12 n (%) | |
| <60% | xx (xx.x%) |
| 60 to 69% | xx (xx.x%) |
| ••• | xx (xx.x%) |
| n | xx |
| Mean Rate | XX.X |
| Median Rate | XX.X |

Table 14.1.7.3 Treatment Adjustments Safety Analysis Set

| Time Period | T | otal |
|---|---|---|
| Exposure Adjustment | ( | N=) |
| Baseline to <week 12<="" td=""><td></td><td></td></week> | | |
| Remained on Istradefyline 20 mg | xx ( | xx.x%) |
| Escalated to Istradefyline 40 mg | xx ( | xx.x%) |
| Escalated to Istradefyline 40 mg and de-escalated to Istradefyline 20 mg | xx ( | xx.x%) |
| Week 12 to <week 26<="" td=""><td></td><td></td></week> | | |
| Remained on Istradefyline 20 mg | xx ( | xx.x%) |
| Remained on Istradefyline 40 mg | xx ( | xx.x%) |
| Escalated to Istradefyline 40 mg | xx ( | xx.x%) |
| Escalated to Istradefyline 40 mg and de-escalated to Istradefyline 20 mg | xx ( | xx.x%) |
| ≥Week 26 | | |
| Remained on Istradefyline 20 mg | xx ( | xx.x%) |
| Remained on Istradefyline 40 mg | xx ( | xx.x%) |
| Total | | |
| Remained on Istradefyline 20 mg (without escalation to 40 mg) | xx ( | xx.x%) |
| Escalated and Remained on Istradefyline 40 mg | xx ( | xx.x%) |
| Escalated to Istradefyline 40 mg and De-escalated to Istradefyline 20 mg | xx ( | xx.x%) |

Note: time period: Baseline to < Week 12, 1 to 84 study days; Week 12 to < Week 26, 85 to 183 study days; ≥ Week 26, ≥ 184 study days

Table 14.2.1.1 Patient Global Impression - Improvement by Study Visit - Overall Condition ITT Analysis Set

Treatment in 6002-014

| | m1 1 | - 1 6 77 1 | |
|---|---|---|---|
| Visit/ | Placebo | Istradefylline | Total |
| Score | (N=) | (N=) | (N=) |
| Week 12 [n(%)] | xx (100%) | xx (100%) | xx (100%) |
| 1=Moderate improvement (or greater) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2=Mild improvement | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3=No change from Baseline | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 4=Mild deterioration | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 5=Moderate deterioration (or greater) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Week 26 [n(%)]

(Note to Programmer: Repeat for week 52)

Kyowa Kirin Pharmaceutical Development, Inc. Istradefylline: Protocol 6002-018

**DDMMMYYYY** Page n of N

Table 14.2.1.2

Patient Global Impression - Improvement by Study Visit - Fatigue ITT Analysis Set

Note to Programmer: Repeat Table 14.2.1.1

Table 14.2.1.3

Patient Global Impression - Improvement by Study Visit - Sleep

ITT Analysis Set

Note to Programmer: Repeat Table 14.2.1.1

Table 14.2.1.4

Patient Global Impression - Improvement by Study Visit - Motivated to Get Things Done

ITT Analysis Set

Note to Programmer: Repeat Table 14.2.1.1

Table 14.2.1.5

Patient Global Impression - Improvement by Study Visit - Key Symptoms

ITT Analysis Set

Note to Programmer: Repeat Table 14.1.5.1
Table 14.3.1.1

Overall Summary of Treatment-Emergent Adverse Events (TEAE)

Safety Analysis Set

| | Total<br>(N=) |
|---------------------------------------------------------|---------------|
| Subjects with any TEAE n (%) | xx (xx.x) |
| Subjects with any serious TEAE n (%) | xx (xx.x) |
| Subjects with any TEAE leading to discontinuation n (%) | xx (xx.x) |
| Subjects with any Related [1] TEAE n (%) | xx (xx.x) |
| Subjects with any Severe TEAE n (%) | xx (xx.x) |
| Subjects who died n (%) | xx (xx.x) |

<sup>[1]</sup> Related = includes probably, possibly, and definitely study drug related.

Table 14.3.1.2

Subjects with Treatment-Emergent Adverse Events (TEAE) by System Organ Class and Preferred Term Safety Analysis Set

| System Organ Class/ | Total |
|------------------------------|-----------|
| Preferred Term | (N=) |
| Subjects with any TEAE n (%) | xx (xx.x) |
| System Organ Class 1 | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) |
| ••• | |
| System Organ Class 2 | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) |
| ••• | |

Programming Notes: For all TEAE tables (where applicable), present the data within an SOC by frequency of occurrence in decreasing order (NOT alphabetically) then by PT within SOC by frequency of occurance.

Same format will be followed for Tables 14.3.1-3, 14.3.1-4.

Table 14.3.1.3
Subjects with Treatment-Emergent Adverse Events (TEAE)
by System Organ Class, Preferred Term, and Maximum Severity
Safety Analysis Set

| | | Total |
|------------------------------------|----------|-----------|
| System Organ Class/ Preferred Term | Severity | (N=) |
| Subjects with any TEAE n (%) | Mild | xx (xx.x) |
| | Moderate | xx (xx.x) |
| | Severe | xx (xx.x) |
| System Organ Class 1 | Mild | xx (xx.x) |
| | Moderate | xx (xx.x) |
| | Severe | xx (xx.x) |
| Preferred Term 1 | Mild | xx (xx.x) |
| | Moderate | xx (xx.x) |
| ••• | Severe | xx (xx.x) |

Note: If a subject experienced more than 1 TEAE within a system organ class, the subject is counted once under that SOC. If a subject has more than 1 count of a particular preferred term, the subject was counted once for that preferred term. If a subject experienced more than 1 severity within a TEAE, the subject is counted once under maximum severity. MedDRA dictionary Version 16.1 was used for coding.

NOTE TO PROGRAMMER: Please present in descending order by total count in SOC, and then in descending order by total count for PT within SOC.

Table 14.3.1.4

Subjects with Treatment-Emergent Adverse Events (TEAE)
by System Organ Class, Preferred Term, and Relationship to Study Drug
Safety Analysis Set

| System Organ Class/ Preferred Term | Relation to Study<br>Drug | Total<br>(N=) |
|---|---|---|
| Subjects with any TEAE n (%) | Related | xx (xx.x) |
| | Not Related | xx (xx.x) |
| System Organ Class 1 | Related | xx (xx.x) |
| | Not Related | xx (xx.x) |
| Preferred Term 1 | Related | xx (xx.x) |
| | Not Related | xx (xx.x) |

Note: If a subject experienced more than 1 TEAE within a system organ class, the subject is counted once under that SOC. If a subject has more than 1 count of a preferred term, the subject was counted once for that preferred term. MedDRA dictionary Version 16.1 was used for coding.

Table 14.3.2.1
Subjects with any Treatment-Emergent Adverse Events Leading to Death by System Organ Class and Preferred Term
Safety Analysis Set

| System Organ Class/ Preferred Term | Total<br>(N=) | Dose at<br>Occurrence | |
|---|---|---|---|
| | , , | 20 mg | 40 mg |
| Subjects with any TEAE leading to death n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ••• | | | |
| System Organ Class 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ••• | | | |

NOTE TO PROGRAMMER: Please present in descending order by frequency in SOC, and then by frequency in descending order by PT within SOC.

Table 14.3.2.2

Subjects with Serious Treatment-Emergent Adverse Events (TEAE) by System Organ Class and Preferred Term Safety Analysis Set

| System Organ Class/<br>Preferred Term | Total<br>(N=) | | Dose at<br>Occurrence |
|---|---|---|---|
| | | 20 mg | 40 mg |
| Subjects with any Serious TEAE n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ••• | | | |
| System Organ Class 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x |
| ••• | | | |

NOTE TO PROGRAMMER: Please present in descending order by frequency in SOC, and then in descending order by frequency PT within SOC.

Table 14.3.2.3

Subjects with Treatment-Emergent Adverse Events (TEAE) Leading to Discontinuation from the Study by System Organ Class and Preferred Term

Safety Analysis Set

| System Organ Class/ Preferred Term | Total (N=) | | Dose at<br>Occurrence |
|---|---|---|---|
| | | 20 mg | 40 mg |
| Subjects with any TEAE Leading to Discontinuation n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ••• | | | |
| System Organ Class 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ••• | | | |

Darameter (IInit)

Table 14.3.4.1

Summary Statistics by Laboratory Test: Hematology
Actual and Change from Baseline Values

Safety Analysis Set

| Total<br>(N=) | |
|---|---|
| Actual C | |
| XX | |
| XX.XX | |
| x.xxx | |
| XX.XX | |
| xx.x-xx.x | |
| XX | XX |
| XX.XX | XX.XX |
| x.xxx | X.XXX |
| XX.XX | XX.XX |
| xx.x-xx.x | xx.x-xx.x |
| | XX XX.XX |

Table 14.3.4.2

Summary Statistics by laboratory Test: Blood Chemistry
Actual and Change from Baseline Values

Safety Analysis Set

Note to Programmer: Repeat Table 14.3.4.1 for Blood Chemistry

Table 14.3.4.3

Summary Statistics by laboratory Test: Urinalysis
Actual and Change from Baseline Values
Safety Analysis Set

Note to Programmer: Repeat Table 14.3.4.1 for Urinalysis

Table 14.3.4.4
Shift Table by Laboratory Test: Hematology
Safety Analysis Set

| | | ourod imario. | | | |
|---|---|---|---|---|---|
| ameter: Hemoglobin (Unit) | | | | | |
| Post-Baseline | | | | | |
| Visit | | | Baseline n ( | (%) | |
| | | High | Low | Normal | Total |
| | High | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x |
| Week 26 | Normal | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x |
| | Low | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x |
| | Total | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | 100% |
| Week 52 | | | | | |
| | High | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x |
| | Normal | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx. |
| | Low | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx. |
| | Total | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | 100% |

Note: High = above upper limit of normal reference range; Normal = within limit of normal reference range; Low = below low limit of normal reference range.

Reference range: see Preface A.

Table 14.3.4.5
Shift Table by Laboratory Test: Blood Chemistry
Safety Analysis Set

Note to Programmer: Repeat Table 14.3.4.4 for Blood Chemistry

Table 14.3.4.6
Shift Table by Laboratory Test: Urinalysis - Continuous Parameters
Safety Analysis Set

Note to Programmer: Repeat Table 14.3.4.4 for Urinalysis - Continuous Parameters

Table 14.3.4.7

Shift Table by Laboratory Test: Urinalysis - Categorical Parameters
Safety Analysis Set

Note to Programmer: Repeat Table 14.3.4.4 for Urinalysis - Categorical Parameters

Listing 16.2.1.1
Subject Completion/Discontinuation

| Clinical | | | | | | |
|---|---|---|---|---|---|---|
| Site | Date of First Dose/ | | Dose at | | | |
| Subject | Date of Last Dose/ | Date/Day of | Final | Completed | Reason for | Analysis |
| No. | Day of Last Dose [1] | Final Visit | Visit (mg) | Study | Discontinuation | Population |
| xxx-xxx | DDMMMYYYY/<br>DDMMMYYYY/XX | DDMMMYYYY/XX | | Yes | | ITT, Safety |
| xxxx-xxx | DDMMMYYYY/<br>DDMMMYYYY/XX | DDMMMYYYY/XX | | No | Adverse Event | ITT, Safety |

Source: Data source: xyzabc.sas7bdat Program source: myprogram.sas

Note to Programmer: Add source to all listings

<sup>[1]</sup> Relative to first dose of study drug.

Listing 16.2.1.2 Screen Failures

Clinical Site

Subject No. Reason for Screen Failure

xxxx-xxx

xxxx-xxx

Source: Data source: xyzabc.sas7bdat Program source: myprogram.sas

Note to Programmer: Add source to all listings

Listing 16.2.2.1
Major Protocol Deviations

| Clinical Site | | Visit Impacted by | |
|---------------|--------------------|-------------------|------------------|
| Subject No. | Protocol Deviation | Deviation | Description |
| XXXX-XXX | | Screening | xxxxxxxxxxxxxxx |
| | | | xxxxxxxxxxxxxxx |
| | | | xxxxxxxxxxxxxxx |
| | | | xxxxxxxxxxxxxxxx |
| | | | xxxxxxxxxxxxxxxx |
| xxxx-xx | | Screening | |

NOTE TO PROGRAMMER: This will be programmed based on data provided by clinical.

Listing 16.2.2.2 Inclusion/Exclusion Criteria Violations

| Clinical Site<br>Subject No | Date of<br>Informed Consent | Satisfy All Eligibility Criteria? | Criteria Not<br>Met | Protocol Subject<br>Initially Consented |
|---|---|---|---|---|
| xxxx-xxx | DDMMMYYYY | No | XX | Amendment 2 |
| xxxx-xxx | DDMMMYYYY | No | I01 E01 | Amendment 3 |
| xxxx-xxx | DDMMMYYYY | No | I02 E05 | Amendment 4 |

# Listing 16.2.3 Subjects Excluded from Analysis Sets

| Clinical Site<br>Subject No. | Analysis Set | Exclusion<br>Yes/No | Reason for Exclusion |
|---|---|---|---|
| xxxx-xxx | ITT | No | |
| | Safety | Yes | xxxxxxxxxxxxxxx |
| xxxx-xxx | ITT | No | |
| | Safety | No | |

Listing 16.2.4.1 Demography

| | | | | | | Smoker/ | | | Of Child- |
|---|---|---|---|---|---|---|---|---|---|
| Clinical | | | | | Height (cm)/ | Cigar- | Caffeine | Number of | Bearing |
| Site | Age | | | | Weight (kg)/ | ettes | Intake | Years of | Potential? |
| Subject No. | (yrs) | Gender | Race | Ethnicity | BMI (kg/m²) | per Day | per Day | Education | |
| xxxx-xxx | XX | Female | XXXX | xxxxxxxxx | xxx.x/ | Yes/<=5 | 2 | 12 Years | Yes/No |
| | | | X | | xx.x/ | / >5 | | | |
| | | | | | XX.X | | | | |
| | XX | Male | XXXX | XXXXXXXXX | XXX.X | No | 1 | >12Years | |
| | | | X | | | | | | |
| xxxx-xxx | | | | | | | | | |
| | XX | Female | XXXX | xxxxxxxxx | XXX.X | No | 3 | >12Years | Yes/No |
| | | | X | | | | | | |
| XXXX-XXX | XX | Male | XXXX | XXXXXXXXX | XXX.X | Yes/xx | 4 | 12Years | |
| | | | X | | | | | | |
| | XX | Male | XXXX | xxxxxxxxx | XXX.X | Yes/xx | | | |
| | | | Х | | | | | | |

### Listing 16.2.4.2 Parkinson's Disease History

| Clinical Site | Linical Site Screening Visit PD Dia | | Levodopa Ir | nitiated | Onset of Motor Complications | |
|---|---|---|---|---|---|---|
| Subject No. | Date/Day [1] | Duration | Date | Duration (Yrs) | Date | Duration (Yrs) |
| xxxx-xxx | DDMMMYYYY/XXX | < 1 year | DDMMMYYYY | XX | DDMMMYYYY | XX |
| xxxx-xxx | DDMMMYYYY/XXX | 1-3 years | DDMMMYYYY | XX | DDMMMYYYY | XX |
| xxxx-xxx | DDMMMYYYY/XXX | 4-7 years | DDMMMYYYY | XX | DDMMMYYYY | XX |

Note: data from Study 6002-014.
[1] Relative to first dose of study drug.

# Listing 16.2.4.3 Medical History

| Subject No. Reported Term Start Date Ongoing? xxxx-xxx XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
|---|
| xxxx-xxx |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

Listing 16.2.4.4.1
Prior Medications (Excluding AntiParkinsonian Medications)

| Clinical Site | Preferred | | Total Daily | Start | Stop | |
|---|---|---|---|---|---|---|
| Subject No. | Term [1] | Medication | Dose (Unit) | Date/Day[2] | Date/Day[2] | Indication |
| xxxx-xxx | XXXXX | XXXXX | 10 mg | DDMMMYYYY/xx | Ongoing | xxxxxxxxx |
| xxx-xxx | xxxxx | xxxxx | 10 mg | DDMMMYYYY/xx | DDMMMYYYY/xx | xxxxxxxxx |
| xxxx-xxx | xxxxx | xxxxx | 10 mg | DDMMMYYYY/xx | DDMMMYYYY/xx | xxxxxxxxx |

<sup>[1]</sup> XXX dictionary Version YYY was used for coding.

<sup>[2]</sup> Relative to first dose of study drug.

Listing 16.2.4.4.2 Concomitant Medications (Excluding AntiParkinsonian Medications)

| Clinical Site | Preferred | | Total Daily | Start | Stop | |
|---|---|---|---|---|---|---|
| Subject No. | Term [1] | Medication | Dose (Unit) | Date/Day[2] | Date/Day[2] | Indication |
| xxxx-xxx | xxxxx | xxxxx | 10 mg | DDMMMYYYY/xx | Ongoing | xxxxxxxxx |
| xxxx-xxx | xxxxx | xxxxx | 10 mg | DDMMMYYYY/xx | DDMMMYYYY/xx | xxxxxxxxx |
| xxxx-xxx | xxxxx | XXXXX | 10 mg | DDMMMYYYY/xx | DDMMMYYYY/xx | xxxxxxxxx |

<sup>[1]</sup> XXX dictionary Version YYY was used for coding.

<sup>[2]</sup> Relative to first dose of study drug.

Listing 16.2.4.5.1 Prior Antiparkinsonian Medications

| Clinical Site | Preferred | | Total Daily | Start | Stop | |
|---|---|---|---|---|---|---|
| Subject No. | Term [1] | Medication | Dose (Unit) | Date/Day[2] | Date/Day[2] | Indication |
| xxxx-xxx | xxxxx | xxxxx | 10 mg | DDMMMYYYY/xx | Ongoing | xxxxxxxxx |
| xxxx-xxx | xxxxx | xxxxx | 10 mg | DDMMMYYYY/xx | DDMMMYYYY/xx | xxxxxxxxx |
| xxxx-xxx | xxxxx | xxxxx | 10 mg | DDMMMYYYY/xx | DDMMMYYYY/xx | xxxxxxxxx |

<sup>[1]</sup> XXX dictionary Version YYY was used for coding.

<sup>[2]</sup> Relative to first dose of study drug.

Listing 16.2.4.5.2 Concomitant Antiparkinsonian Medications

| Clinical Site | Preferred | | Total Daily | Start | Stop | |
|---|---|---|---|---|---|---|
| Subject No. | Term [1] | Medication | Dose (Unit) | Date/Day[2] | Date/Day[2] | Indication |
| xxxx-xxx | XXXXX | xxxxx | 10 mg | DDMMMYYYY/xx | Ongoing | xxxxxxxxx |
| xxxx-xxx | xxxxx | xxxxx | 10 mg | DDMMMYYYY/xx | DDMMMYYYY/xx | xxxxxxxxx |
| xxxx-xxx | xxxxx | xxxxx | 10 mg | DDMMMYYYY/xx | DDMMMYYYY/xx | xxxxxxxx |

<sup>[1]</sup> XXX dictionary Version YYY was used for coding.

<sup>[2]</sup> Relative to first dose of study drug.

Listing 16.2.5.1 Study Drug Dosing Record and Compliance

| Clinical<br>Site | | | | | Number of<br>Tablets | Number of<br>Tablets | | 70% or<br>Greater | Reason for |
|---|---|---|---|---|---|---|---|---|---|
| Subject | | Date Dispensed-day/ | Bottle | Dose | Dispensed | Returned | Compliance | Compl- | Non- |
| No. | Visit | Returned-day [1] | Number | Level | 40 mg/20mg | 40mg/20mg | Rate [2] | iant? | compliance |
| xxxx-xxx | xxx | DDMMMYYYY-xx/<br>DDMMMYYYY-xx | XXX | 20 mg/d | xxx/xxx | xxx/xxx | xx.x% | No | AE |
| xxxx-xxx | XXX | DDMMMYYYY-xx/<br>DDMMMYYYY-xx | xxx | 40 mg/d | xxx/xxx | xxx/xxx | xx.x% | No | Other:XXXX |
| xxxx-xxx | XXX | DDMMMYYYY-xx/<br>DDMMMYYYY-xx | xxx | 20 mg/d | xxx/xxx | xxx/xxx | xx.x% | Yes | |

#### Note:

<sup>[1]</sup> Relative to first dose of study drug.
[2] Compliance rate = [(Number of tablets dispensed - Number of tablets returned) / (Number of tablets expected to be taken)] \* 100.

### Listing 16.2.5.2 Study Drug Dose Adjustment

| Clinical<br>Site | | Assessment | Was the Dose<br>Level | Reason for Dose | | If Other, |
|---|---|---|---|---|---|---|
| Subject No. | Visit | Date/Day [1] | Adjusted? | Adjustment | If AE, Specify | specify |
| xxxx-xxx | xxx | DDMMMYYYY/XX | Yes | xxxxxxxxx | xxxxxxxxx | xxxxxxxxxx |
| xxx-xxx | xxx | DDMMMYYYY/XX | No | | | |
| xxxx-xxx | XXX | DDMMMYYYY/XX | No | | | |

#### Note:

[1] Relative to first dose of study drug.

Listing 16.2.6
Patient Global Impression - Improvement

| Clinical Site Subject No. | Visit | Assessment Date/Day [1] | Overall<br>Condition<br>[2] | Fatigue<br>[2] | Sleep [2] | Motivated<br>to Get<br>Tasks Done<br>[2] | Key Symptom |
|---|---|---|---|---|---|---|---|
| xxxx-xxx | End of 6002-014 | DDMMMYYYY/XX | | | | | XXXXXXX/4 |
| | Baseline | DDMMMYYYY/XX | | | | | XXXXXXX/5 |
| | Week 12 | DDMMMYYYY/XX | 1 | 2 | 3 | 4 | XXXXXXX/5 |
| | Week 26 | DDMMMYYYY/XX | 1 | 2 | 3 | 4 | XXXXXXX/5 |
| | Week 52 | DDMMMYYYY/XX | 1 | 2 | 3 | 4 | XXXXXXX/5 |
| xxxx-xxx | End of 6002-014<br>Baseline | DDMMMYYYY/XX<br>DDMMMYYYY/XX | | | | | XXXXXXX/4<br>XXXXXXX/3 |
| | Week 12 | DDMMMYYYY/XX | 1 | 2 | 3 | 4 | XXXXXXX/3 |

<sup>[1]</sup> Relative to first dose of study drug.

<sup>[2]</sup> PGI-I Scale: 1=Moderate improvement (or greater), 2=Mild improvement, 3=No change from Baseline, 4=Mild deterioration, 5=Moderate deterioration (or greater).

Listing 16.2.7.1 Adverse Events

| | | AE Start | AE Stop | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Clinical | | | | Istra- | | | | | |
| Site | | | | defylline | | | | Action | |
| Subject | | Date/ | Date/ | dose at | | Severity | Relation | taken | Outcome |
| No. | SOC/PT/Verbatim | Day [1] | Day [1] | AE onset | SAE | [2] | [3] | [4] | [5] |
| | | | | | | | Def/ | Drug | Res/ |
| | | | | | | | Prob/ | W/D/ | Res'ing/ |
| | | | | | | | Poss/ | Dose | Not Res/ |
| | XXXXXXXX | | | | | Mild/ | Unlike/ | Int/ | Res Seq/ |
| | /xxxxxxxxx | DDMMMYYYY/ | DDMMMYYYY/ | | | Mod/ | Not R/ | No Chg; | Fatal/ |
| XXXX | /xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XX | XX | | Yes | Severe | N/A | N/A | Unk |

Note: XXX dictionary Version YYY was used for coding. AE=Adverse Event; SOC=System Organ Class; PT=Preferred Term; SAE=Serious Adverse Event.

- [1] Relative to first dose of study drug. Negative days at AE Start indicate the AE occured prior to first dose.
- [2] Severity: Mod=Moderate.
- [3] Relationship to Study Drug: Def=Definitely; Prob=Probably; Poss=Possibly; Unlike=Unlikely; Not R=Not Related; N/A=Not Applicable.
- [4] Action taken: Drug W/D=Drug Withdrawn; Dose Int=Dose Interrupted; No Chg=Dose Not Changed; N/A=Not Applicable.
- [5] Outcome: Res=Recovered/Resolved; Res'ing=Recovering/Resolving; Not Res=Not Recovered/Not Resolved; Res Seq= Recovered/Resolved with Sequelae; Unk=Unknown.

### Listing 16.2.7.2 Serious Adverse Events and Deaths

| | | AE Start | AE Stop | | | | | |
|---|---|---|---|---|---|---|---|---|
| Clinical | | | | Istra- | | | | |
| Site | | | | defylline | Sever- | | Action | |
| Subject | | Date/ | Date/ | dose at AE | ity | Relation | taken | Outcome |
| No. | SOC/PT/Verbatim | Day [1] | Day [1] | onset | [2] | [3] | [4] | [5] |
| | | | | | | Def/ | Drug | Res/ |
| | | | | | | Prob/ | W/D/ | Res'ing/ |
| | | | | | | Poss/ | Dose | Not Res/ |
| | XXXXXXXX | | | | Mild/ | Unlike/ | Int/ | Res Seq/ |
| | /xxxxxxxxxx | DDMMMYYYY/ | DDMMMYYYY/ | | Mod/ | Not R/ | No Chg; | Fatal/ |
| XXXX | /xxxxxxxxxxxxxx | XX | XX | | Severe | N/A | N/A | Unk |

Note: XXX dictionary Version YYY was used for coding. AE=Adverse Event; SOC=System Organ Class; PT=Preferred Term; SAE=Serious Adverse Event.

- [1] Relative to first dose of study drug. Negative days at AE Start indicate the AE occured prior to first dose.
- [2] Severity: Mod=Moderate.
- [3] Relationship to Study Drug: Def=Definitely; Prob=Probably; Poss=Possibly; Unlike=Unlikely; Not R=Not Related; N/A=Not Applicable.
- [4] Action taken: Drug W/D=Drug Withdrawn; Dose Int=Dose Interrupted; No Chg=Dose Not Changed; N/A=Not Applicable.
- [5] Outcome: Res=Recovered/Resolved; Res'ing=Recovering/Resolving; Not Res=Not Recovered/Not Resolved; Res Seq= Recovered/Resolved with Sequelae; Unk=Unknown.

Kyowa Kirin Pharmaceutical Development, Inc. Istradefylline: Protocol 6002-018

DDMMMYYYY Page n of N

Listing 16.2.7.3

Adverse Events Leading to Discontinuation from the Study

Note to Programmer: Repeat listing 16.2.7.1 for AE Leading to Discontinuation from the Study.

Listing 16.2.8.1 Laboratory Assessments - Hematology

| Clinical | | | | | | | |
|---|---|---|---|---|---|---|---|
| Site<br>Subject No. | Parameter | Unit | Normal Range<br>Low-High | Visit | <pre>Sample Date/Time/Day [1]</pre> | Lab Value | Flag* |
| XXX-XXX | xxxxxxxxxxxxxx | XXX | xx.x - xx.x | XXXXXXX | DDMMMYYYY/HH:MM/XXX | XX.X | |
| | | | | XXXXXXX | DDMMMYYYY/HH:MM/XXX | XX.X | H |
| | | | | xxxxxxx | DDMMMYYYY/HH:MM/XXX | XX.X | |
| | xxxxxxxxxxxx | XXX | xx.x - xx.x | xxxxxxx | DDMMMYYYY/HH:MM/XXX | xx.x | |
| | | | | XXXXXXX | DDMMMYYYY/HH:MM/XXX | XX.X | Н |
| | | | | xxxxxxx | DDMMMYYYY/HH:MM/XXX | XX.X | |
| | xxxxxxxxxxxxxx | xxx | xx.x - xx.x | xxxxxxx | DDMMMYYYY/HH:MM/XXX | xx.x | |
| | | | | XXXXXXX | DDMMMYYYY/HH:MM/XXX | XX.X | Н |
| | | | | xxxxxxx | DDMMMYYYY/HH:MM/XXX | XX.X | |
| xxx-xxx | xxxxxxxxxxxx | XXX | xx.x - xx.x | xxxxxxx | DDMMMYYYY/HH:MM/XXX | XX.X | |
| ANA ANA | MAMAMAMAMAMA | 22222 | AA.A AA.A | XXXXXXXX | DDMMMYYYY/HH:MM/XXX | XX.X | Н |
| | | | | xxxxxxx | DDIMITITITY IIII (IIII) | 222. | |
| | xxxxxxxxxxxxx | xxx | xx.x - xx.x | xxxxxxx | DDMMMYYYY/HH:MM/XXX | XX.X | |
| | | | | XXXXXXX | DDMMMYYYY/HH:MM/XXX | XX.X | Н |
| | | | | xxxxxxx | DDMMMYYYY/HH:MM/XXX | XX.X | |
| xxx-xxx | xxxxxxxxxxxx | XXX | xx.x - xx.x | xxxxxxx | DDMMMYYYY/HH:MM/XXX | XX.X | |
| | | | | XXXXXXX | DDMMMYYYY/HH:MM/XXX | XX.X | Н |

65

Note: CS = clinically significant.
[1] Relative to first dose of study drug.

<sup>\*</sup> H = above upper limit of normal reference range; L = below lower limit of normal reference range.

Kyowa Kirin Pharmaceutical Development, Inc. Istradefylline: Protocol 6002-018

DDMMMYYYY Page n of N

Listing 16.2.8.2 Laboratory Assessments - Blood Chemistry

Note to Programmer: Repeat listing 16.2.8.1 for blood chemistry parameters

Listing 16.2.8.3 Laboratory Assessments - Urinalysis

Note to Programmer: Repeat listing 16.2.8.1 for urinalysis parameters

Listing 16.2.8.4 Pregnancy Test

| Clinical Site | | Assessment | | |
|---------------|-----------|---------------|-------------|----------|
| Subject No. | Visit | Date/Day [] | Sample Type | Result |
| xxxx-xxx | Screening | DDMMMYYYY/XXX | Serum | Negative |
| | Day 1 | DDMMMYYYY/XXX | Urine | Negative |
| | Week 26 | DDMMMYYYY/XXX | Serum | Negative |
| | Week 52 | DDMMMYYYY/XXX | Serum | Negative |
| xxxx-xxx | Screening | DDMMMYYYY/XXX | Serum | Negative |
| | Day 1 | DDMMMYYYY/XXX | Urine | Negative |

<sup>[1]</sup> Relative to first dose of study drug.

# Listing 16.2.8.5 Follicle Stimulating Hormone

| Clinical Site | | Assessment Date/Day | Assessment Date/Day |
|---|---|---|---|
| Subject No. | Visit | [1] | FSH > 30 IU/L |
| XXXX-XXX | Screening | DDMMMYYYY/XX | Yes |

<sup>[1]</sup> Relative to first dose of study drug.

### Listing 16.2.8.6 Laboratory Assessments - Comments

| Clinical<br>Site | | Normal<br>Range | | Sample Date/Day | ate/Day Lab | |
|---|---|---|---|---|---|---|
| Subject No. | Parameter (Unit) | Low-High | Visit | [1]/Time | Value | Comment |
| xxx-xxxxxx | xxxxxxx (xxxxxx) | x.x-x.x | Week xx | ddMMMyyyy/xx/hh:mm | х.х | <text></text> |
| | xxxxxxx (xxxxxx) | x.x-x.x | Week xx<br>Week xx | ddMMMyyyy/xx/hh:mm<br>ddMMMyyyy/xx/hh:mm | x.x<br>x.x | <text><br/><text></text></text> |

(Programming Note:Only list lab data having an associated comment in SDTM dataset SUPPLB.)

Listing 16.2.9.1 Vital Signs and Body Weight

| Clinical Site Subject No. | Visit | Assessment Date/Day [1] | Height<br>(cm) | Weight<br>(kg) | Systolic<br>BP<br>(mmHg) | Diastolic<br>BP (mmHg) | Heart<br>Rate<br>(bpm) | Respiratory<br>Rate<br>(resp/min) | Temp<br>(C) |
|---|---|---|---|---|---|---|---|---|---|
| xxxx-xxx | Screening | DDMMMYYYY/<br>XX | XXX | XXX | XXX | XXX | XXX | XX | XX.X |
| | Unscheduled | DDMMMYYYY/XX | | | | | | XX | XX.X |
| xxxx-xxx | Screening | DDMMMYYYY/XX | | | | | | | |
| | Unscheduled | DDMMMYYYY/XX | | | | | | | |

Note: Height was only collected at screening. Only screening systolic/diastolic blood pressure and heart rate are presented on this listing..

[1] Relative to first dose of study drug.

### Listing 16.2.9.2 12-Lead Electrocardiogram Report - Qualitative Data by Subject

| Clinical Site Subject No. Visit | | Assessment Date/Day | Assessment Date/Day [1] Assessment Time | |
|---|---|---|---|---|
| xxxx-xxx | Screening | DDMMMYYYY/XX | TIOGESOMETIC TIME | Result [2] |
| | Unscheduled | DDMMMYYYY/XX | XX:XX | Abnormal, CS |
| xxxx-xxx | Screening | DDMMMYYYY/XX | | |
| | Unscheduled | DDMMMYYYY/XX | XX:XX | Abnormal, CS |

<sup>[1]</sup> Relative to first dose of study drug.

<sup>[2]</sup> CS=Clinically significant.

## Listing 16.2.9.3 Physical Examination

| Clinical Site Subject No. | Visit | Assessment Date/Day [1] | Assessment Time | Physical Exam<br>Findings [2] |
|---|---|---|---|---|
| Subject No. | | * | Assessment rime | FINALINGS [2] |
| xxxx-xxx | Screening | DDMMMYYYY/XX | | |
| | Unscheduled | DDMMMYYYY/XX | | |
| xxxx-xxx | Screening | DDMMMYYYY/XX | | |
| | Unscheduled | DDMMMYYYY/XX | | |

<sup>[1]</sup> Relative to first dose of study drug.

<sup>[2]</sup> CS=Clinically significant.

# Listing 16.2.9.4 Neurological Examination

| linical Site | | | | Neurological Exam |
|---|---|---|---|---|
| Subject No. | Visit | Assessment Date/Day [1] | Assessment Time | Findings [2] |
| xxxx-xxx | Screening | DDMMMYYYY/XX | XX:XX | Normal |
| | Unscheduled | DDMMMYYYY/XX | | |
| xxxx-xxx | Screening | DDMMMYYYY/XX | | |
| | Unscheduled | DDMMMYYYY/XX | | |

73

<sup>[1]</sup> Relative to first dose of study drug.

<sup>[2]</sup> CS=Clinically significant.